CLINICAL TRIAL: NCT03123536
Title: Effects of Perioperative Point-of-care Ultrasound Assessment on Postoperative Outcomes in High Risk Surgical Patients
Brief Title: Use of Point-of-care Ultrasound in High Risk Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jian-jun Yang, Director, Department of Anesthesiology, Zhongda Hospital
Other Study IDs: 20161226
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Ultrasonography; Outcomes; Cardiopulmonary
Keywords: high risk; complication; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Point-of-care ultrasound group: High risk patients received point-of-care ultrasound assessment perioperatively, treatment was oriented by the findings of point-of-care ultrasound.
  Interventions: Device: Point-of-care Ultrasound
- Control group: High risk patients received management by the experience of the clinical team.

INTERVENTIONS:
Device: Point-of-care Ultrasound — Patients' management in the point-of-care ultrasound group will be adjusted according to the results of ultrasound, whereas patients in the control group the decisions about the management were made by the experience of clinical team.
  Groups: Point-of-care ultrasound group

SUMMARY:
There is currently a lack of evidence to support the use of perioperative point-of-care ultrasound to assess the outcomes in high risk surgical patients. Thus, the purposes of this study were to evaluate whether perioperative use of point-of-care ultrasound can reduce the worse postoperative outcomes in high surgical patients.

DETAILED DESCRIPTION:
Point-of-care ultrasound is increasingly established as a useful bedside tool when performed by the anesthesiologist for evaluation of cardiopulmonary dysfunction and other emergent situations. However, it remains unclear whether use of perioperative point-of-care ultrasound can reduce the worse postoperative outcomes in high surgical risk patients.

Patients were randomly allocated to two groups. In the point-of-care ultrasound group, treatment was oriented by the findings of point-of-care ultrasound, while in the control group the decisions about the management of patients were made by the experience of the clinical team. The primary outcome measures were hospital mortality and 28-day mortality, and the secondary outcome measures were the complications and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have comprised cardiovascular，respiratory diseases，or other critical illness.

Exclusion Criteria:

* Patients who decline to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: More and more high risk patients undergo surgery,which is associated with increased morbidity and mortality. The aim of the present study was to investigate the value of point-of-care ultrasound for assessment of postoperative outcomes in high risk surgical patients.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Hypotension | Within 7 days after surgery
  Patients who have hypotension which is defined by mean arterial pressure less than 60 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No